CLINICAL TRIAL: NCT01144260
Title: A Pilot Phase II Study of Bafetinib (INNO-406) as Treatment for Patients With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Study of Bafetinib as Treatment for Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAFETINIB-P2-CLL-01
Record Dates: First submitted 2010-06-09; First posted 2010-06-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: CLL; leukemia; chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — bafetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bafetinib (Experimental)
  Interventions: Drug: bafetinib

INTERVENTIONS:
Drug: bafetinib — 250 mg orally twice daily. Treatment continues until clinically significant disease progression or unacceptable toxicity is documented.
  Other Names: INNO-406

SUMMARY:
A Study of Bafetinib as Treatment for Patients with Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia (B-CLL).

DETAILED DESCRIPTION:
Bafetinib is a dual protein kinase inhibitor, targeting both bcr/abl and Lyn kinases. B-cell chronic lymphocytic leukemia cells overexpress Lyn kinase compared to normal B lymphocytes as well as acute leukemias (ALL and AML), and inhibition of Lyn kinase induces apoptosis in cultures of B-CLL cells. Thus, bafetinib may stop the growth of B-CLL cells by inhibiting Lyn kinase, the molecule that couples the B cell receptor to downstream signaling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, male or female.
* B-cell chronic lymphocytic leukemia meeting the WHO criteria.
* Relapsed or refractory disease with at least one of the following criteria: *progression after at least one course of a purine nucleoside analog (fludarabine phosphate, cladribine, pentostatin)

  * progression after at least one course of an alkylating agent (cyclophosphamide or chlorambucil)
  * relapse within 12 months after at least one course of either a purine nucleoside or an alkylating agent.
* Capable of providing informed consent and complying with trial procedures.
* ECOG performance status 0-2.
* Requires chemotherapy for disease as shown by any of the following criteria:

  * measurable and progressive lymphocytosis
  * measurable and progressive lymphadenopathy (lymph node ≥2 cm in a single diameter)
  * either weight loss ≥10% within the past 6 months or extreme fatigue due to leukemia
  * fevers ≥100.5 degrees F for 2 weeks with no source of infection
  * night sweats with no evidence of infection
  * progressive marrow failure (worsening anemia with hemoglobin <10 gm/dL and/or thrombocytopenia with platelet count <100,000/mm3)
  * massive or progressive splenomegaly (spleen >6 cm below left costal margin).
* Women must not be able to become pregnant (e.g. post menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. [Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.]
* Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
* Accessibility to the site.

Exclusion Criteria:

* Chemotherapy, antibody therapy, surgery within 4 weeks of study enrollment.
* Exposure to any investigational agent within 30 days of the Screening Visit.
* Known CNS disease.
* Concurrent active malignancies except basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix.
* Laboratory values: Screening creatinine clearance (calculated by Cockcroft Gault formula) of less than 50 mL/minute, alanine aminotransferase (ALT) greater than 3 times the upper limit of normal, total bilirubin greater than 3 times the upper limit of normal, white blood cell (WBC) count <3500/mm3, absolute neutrophil count <1000/mm3, hematocrit level <33% for females or <35% for males.
* Clinically evident congestive heart failure >class II of the New York Heart Association (NYHA) guidelines.
* Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* History or signs of active coronary artery disease with or without angina pectoris.
* Serious myocardial dysfunction defined scintigraphically (MUGA, myocardial scintigram) or ultrasound determined absolute left ventricular ejection fraction (LVEF) <45% of predicted.
* Known HIV infection.
* Uncontrolled active, infection.
* Major surgery within 3 weeks prior to treatment.
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
* Any condition that in the opinion of the Investigator is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate (complete and partial), in subjects with relapsed or refractory B-Cell CLL | Upto 6 months or disease progression

SECONDARY OUTCOMES:
Adverse Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Levitt, M.D., Ph.D., Study Director — CytRx
Locations (2):
- United States (2):
  - City of Hope National Medical Center, Duarte, California
  - UT M.D. Anderson Cancer Center, Houston, Texas